CLINICAL TRIAL: NCT06524024
Title: Clinical Study of Tumor Polypeptide DC-CTL in the Treatment of Solid Tumors
Acronym: DC-CTL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou Revo-Gene Technology Co., LTD (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG2401
Record Dates: First submitted 2024-07-16; First posted 2024-07-29 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Biological: DC-CTL DC combined with CTL
  Interventions: Biological: Tumor polypeptide pool induced DC-CTL cell injection

INTERVENTIONS:
Biological: Tumor polypeptide pool induced DC-CTL cell injection — In this study, DC-CTL cells were injected once a day for two consecutive days, 1-2 days after study participants received a conventional antitumor regimen, and subcutaneous injections of DC cells were administered before a second infusion of DC-CTL cells. A total of about 4-6 cycles of cell infusion are required

SUMMARY:
This clinical study is a real-world exploratory study to observe the safety and initial effectiveness of DC-CTL cells combined with conventional anti-tumor therapy in patients with colorectal cancer, esophageal cancer, lung cancer, liver cancer, breast cancer and other solid tumors.

DETAILED DESCRIPTION:
This clinical study is a real-world exploratory study to observe the safety and initial effectiveness of DC-CTL cells combined with conventional anti-tumor therapy in patients with colorectal cancer, esophageal cancer, lung cancer, liver cancer, breast cancer and other solid tumors. In this study, DC-CTL cells were injected once a day for two consecutive days, 1-2 days after study participants received a conventional antitumor regimen, and subcutaneous injections of DC cells were administered before a second infusion of DC-CTL cells. A total of about 4-6 cycles of cell infusion are required, and the specific number of infusion and the composition of the peptide pool are determined by the investigator based on clinical needs and test results. After the cells have been transfused, their safety is examined first, and their effectiveness is evaluated during follow-up. According to the needs, this study plans to enroll about 20-200 patients with solid tumors such as colorectal cancer, esophageal cancer, lung cancer, liver cancer, and breast cancer. If the disease progresses during treatment, it is evaluated comprehensively by the investigator according to the clinical situation to determine whether the patient can be withdrawn from the study. Study participants in the follow-up phase who develop disease progression, begin other anti-tumor therapy without reaching disease progression after infusion, and voluntarily request to withdraw from the follow-up phase will be withdrawn from the follow-up phase and will be followed for survival only.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Patients clinically diagnosed with solid tumors such as colorectal cancer, esophageal cancer, lung cancer, liver cancer, breast cancer, etc., who need routine anti-tumor therapy;
3. KPS score ≥80 (Appendix 1), expected survival ≥3 months;
4. If imaging is available, the target lesion can be measured by conventional CT or MRI≥10 mm, and the short diameter of lymph node ≥15mm;
5. Liver function: TBIL≤3ULN, AST, ALT ≤2.5ULN; Renal function: Cr≤1.25ULN; Blood routine: WBC ≥ 4.0×109/L, Hb ≥90 g/L, PLT ≥ 80×109/L;
6. Good cardiac function (LVEF≥ 50%);
7. The peripheral superficial veins of the study participants were smooth, which could meet the needs of intravenous infusion;
8. No history of other malignant tumors, except for cured carcinoma in situ and papillary thyroid carcinoma;
9. Study participants agree to use a reliable contraceptive method for contraception from the time of signing the informed consent to the entire clinical study;
10. Study participants agree to participate in the clinical study and sign the Informed Consent form.

Exclusion Criteria:

1. Pregnant or lactating women (women of childbearing age need to do pregnancy tests);
2. Had a serious, uncontrolled infectious disease (bacterial, viral, or fungal infection) within 4 weeks prior to enrollment;
3. have chronic active hepatitis, AIDS or syphilis;
4. have a serious autoimmune disease or immunodeficiency disease (such as systemic lupus erythematosus, inflammatory bowel disease, multiple sclerosis, rheumatoid arthritis, psoriasis);
5. Severe allergy;
6. serious mental disorders;
7. suffering from serious heart, liver, kidney dysfunction, serious uncontrollable diabetes and other diseases;
8. Patients who had systematically used large amounts of glucocorticoids in the 4 weeks prior to enrollment (except those who used inhaled hormones);
9. Those who have previously been treated with other gene products;
10. Other investigators consider it inappropriate to participate in the study, or other circumstances that affect the analysis of the results of this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-11 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From the time of the first cell transfusion to the time of the subject's death due to any cause, up to 2 years after the subject received the last treatment
  progression free survival time

SECONDARY OUTCOMES:
OS | From the time of the first cell transfusion to the time of the subject's death due to any cause, up to 2 years after the subject received the last treatment
  over all survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, professor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No